CLINICAL TRIAL: NCT04839536
Title: A Comparative Study of Sevoflurane Sedation With TCI Propofol Sedation in Dialysis Dependent End Stage Renal Failure Patients for Transposition of Brachiocephalic Fistula Repair
Brief Title: Comparing Sevoflurane With Propofol Sedation in ESRF Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MREC: 2021116-9722
Record Dates: First submitted 2021-03-28; First posted 2021-04-09 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Sevoflurane; Kidney Diseases; Procedural Hypotension
Keywords: Sevoflurane Sedation, ESRF
MeSH Terms: conditions — Kidney Diseases | interventions — Sevoflurane

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Target controlled infusion (TCI) propofol (Active Comparator): For TCI propofol group, all patients will receive nasal CPAP mask and nasal breathing with oxygen of 3 litre/min. We will utilize the Schneider model to target effect-site (Cet) starting from 0.5 mcg/ml and with a gradual 0.5mcg/ml increment every 30s until OAAS score of 3 is achieved. For any patients with OAAS score < 3, Cet will be decreased by a decremental 0.5 mcg/ml. The deepest level of sedation will be recorded.
  Interventions: Drug: Sevoflurane inhalant product
- Sevoflurane sedation (Experimental): Patients randomised to this arm will be given time to familiarise with the nasal continuous positive airway pressure (CPAP) mask and nasal breathing with oxygen 3 litre/min via a Bain anaesthetic circuit before the introduction of sevoflurane. Once the patient starts to adapt to nasal CPAP mask, sevoflurane will be delivered, starting with a concentration of 0.2% and increase stepwise by 0.2% every 30s until sedation score of OAAS of 3 is achieved. Anaesthetist in charge will assess and maintain sedation endpoint to OAAS 3. If patient is over sedated, sevoflurane concentration will be reduced by 0.2% until OAAS 3. The deepest level of sedation will be recorded.
  Interventions: Drug: Sevoflurane inhalant product

INTERVENTIONS:
Drug: Sevoflurane inhalant product — Sevoflurane will be delivered in an incremental dose to throughout procedure to achieve clinical sedation endpoint OAAS 3.
  Other Names: Ultane, 74412392

SUMMARY:
End-stage renal failure (ESRF) cohorts undergo brachiocephalic fistula(BCF) transposition with supraclavicular block. However, this is inadequate because the incision may extend to the axillary region which requires intercostobrachial (T2) dermatome blockage. Sedation is commonly indicated to allay anxiety whilst allowing intraprocedural lignocaine infiltration. It is challenging to administer safe sedation to ESRF patients due to multiple comorbidities, polypharmacy, altered pharmacokinetic drug handling. Intraoperative hypotension can be common and evident from the residual effect of antihypertensive and intravascular hypovolemia from regular hemodialysis. Midazolam is metabolized to an active metabolite which can accumulate causes apnea and delayed recovery. TCI propofol needs higher induction doses to achieve hypnosis causes exaggerated hypotension which may jeopardize organ perfusion. The investigators are exploring the potential benefit of sevoflurane sedation which are independent of renal clearance, rapid onset and offset, and ischemic preconditioning property in ESRF cohorts.

DETAILED DESCRIPTION:
Regional anesthesia has been shown to be superior to general anesthesia in end-stage renal disease (ESRF) patients undergoing brachiocephalic transposition by ensuring graft patency, reducing pharmacokinetic (pK) and pharmacodynamic (pD) unpredictability, and minimize hemodynamic instability. However, a supraclavicular nerve block is inadequate in BCF transposition where surgical incision may extend to the axillary region which requires intercostobrachial nerve (T2) dermatome to be blocked. Intraprocedural lignocaine infiltration or pectoralis minor (PEC 2) block may be required to anaesthetize this region. Hence, sedation is commonly indicated to allay anxiety and to blunt sympathetic stress response to surgery.

ESRF patient is a challenging cohort to administer safe sedation due to multiple comorbidities, polypharmacy, altered pK handling of drug with a high proportion of total body water, the altered volume of distribution, protein binding, drug metabolism and excretion[3]. Commonly used intravenous midazolam causes delayed recovery and apnoea due to loss of renal ability to clear active metabolite α1-hydroxymidazolam. Target controlled infusion (TCI) propofol needs a higher induction dose to achieve clinical end-point of hypnosis in ESRF patient and causes hemodynamic disturbances.

Dialysis dependent ESRF patients are commonly hypertensive and adapted to a higher baseline blood pressure. Intraoperative hypotension is exaggerated from residual effect of antihypertensive, relative intravascular hypovolemia from pre-op haemodialysis and pre-operative fasting with no replacement fluid. Blood pressure determine perfusion, and existing evidence suggests intraoperative hypotension is associated with stroke, myocardial injury and delirium. Major hypertension guidelines have recommended target blood pressure level of 140/90 mm Hg for patients with renal disease.

Volatile sedation with sevoflurane in intensive care has been widely appraised for significant shorten and superior awakening time and reduced incidence of delirium compared with conventional midazolam/ propofol intravenous sedation. Sevoflurane has rapid onset of action with no significant concern of tolerance and tachyphylaxis. Drug clearance is via pulmonary exhalation which is independent of hepatic and renal function. Volatile agent is a mild analgesia with opioid sparing effect via N methyl-D-aspartate receptor blockade, thus provide a more stable sedation profile.ESRF patients are prone to develop ischemic heart disease due to calcification of intima. Sevoflurane also possess ischemic preconditioning and end organ cytoprotective properties along with anti-inflammatory mechanism.

ELIGIBILITY:
Inclusion Criteria:

* Patient with end stage renal failure, dialysis dependent undergoing transposition of brachiocephalic fistula repair
* American Society of Anesthesiology Physical Status Classification System (ASA) II or III

Exclusion Criteria:

* Patient refusal
* History or family history of malignant hyperthermia
* Known allergy to propofol or local anaesthetic agent
* Patients who have taken neuroleptics, benzodiazepine over 2 weeks within 1 month
* Chronic use of alcohols/ opioid
* Active lungs disease (eg. acute exacerbation of chronic obstructive pulmonary disease)
* Active and significant cardiac disease (eg. decompensated congestive cardiac failure, recent myocardial infarction)
* End-stage heart failure with left ventricular ejection fraction < 30%
* Recent (< 3 months) cerebrovascular accident

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in mean arterial pressure from baseline following sedation | At baseline, pre-, and immediately after intervention
  Hemodynamic instability is defined as event below:
  Hypotension- Drop in mean arterial pressure (MAP) from baseline by more than 20% Hypotension - Drop in systolic blood pressure (sBP < 140 mmHg) and diastolic blood pressure (dBP < 90 mmHg)

SECONDARY OUTCOMES:
Number of hemodynamic interventions required during sedation | At baseline, pre-, and immediately after intervention
  administration of vasoactive drugs to maintain hemodynamic within target (sBP> 140 mmHg, dBP > 80 mmHg, MAP within 20% baseline)
Duration of hemodynamic instability | At baseline, pre-, and immediately after intervention and surgery
  Time course of drop in mean arterial pressure more than 20%
Onset time and recovery time | At baseline, pre-, and immediately after intervention and surgery
  Onset time: time from starting sedation to Observer Assessment of Alertness/ Sedation (OAAS) score 3 (maintain at 3 for a consecutive 15 mins) Recovery time: Time from cessation of sedation to return to OAAS score 5

CONTACTS AND LOCATIONS:
Overall Officials: Chao Chia Cheong, MMed Master, Principal Investigator — University of Malaya

IPD SHARING:
Plan to Share IPD: Yes
All collected individual participant data (IPD) and all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Starting 6 months after publication
Access Criteria: Personal enquiry via email

REFERENCES:
- [Background] Quek KH, Low EY, Tan YR, Ong ASC, Tang TY, Kam JW, Kiew ASC. Adding a PECS II block for proximal arm arteriovenous access - a randomised study. Acta Anaesthesiol Scand. 2018 May;62(5):677-686. doi: 10.1111/aas.13073. Epub 2018 Jan 22. PMID 29359313
- [Background] Rutkowska K, Knapik P, Misiolek H. The effect of dexmedetomidine sedation on brachial plexus block in patients with end-stage renal disease. Eur J Anaesthesiol. 2009 Oct;26(10):851-5. doi: 10.1097/EJA.0b013e32832a2244. PMID 19550340
- [Background] Virmani S, Onuchic A, El-Ali IM, Trivedi RD. Propofol Induced Hyperkalemia and Its Management in End Stage Renal Disease Patients. Conn Med. 2016 Sep;80(8):491-493. PMID 29782787
- [Background] Zhong W, Zhang Y, Zhang MZ, Huang XH, Li Y, Li R, Liu QW. Pharmacokinetics of dexmedetomidine administered to patients with end-stage renal failure and secondary hyperparathyroidism undergoing general anaesthesia. J Clin Pharm Ther. 2018 Jun;43(3):414-421. doi: 10.1111/jcpt.12652. Epub 2017 Dec 16. PMID 29247451
- [Background] Xie X, Atkins E, Lv J, Bennett A, Neal B, Ninomiya T, Woodward M, MacMahon S, Turnbull F, Hillis GS, Chalmers J, Mant J, Salam A, Rahimi K, Perkovic V, Rodgers A. Effects of intensive blood pressure lowering on cardiovascular and renal outcomes: updated systematic review and meta-analysis. Lancet. 2016 Jan 30;387(10017):435-43. doi: 10.1016/S0140-6736(15)00805-3. Epub 2015 Nov 7. PMID 26559744
- [Background] Maheshwari K, Ahuja S, Khanna AK, Mao G, Perez-Protto S, Farag E, Turan A, Kurz A, Sessler DI. Association Between Perioperative Hypotension and Delirium in Postoperative Critically Ill Patients: A Retrospective Cohort Analysis. Anesth Analg. 2020 Mar;130(3):636-643. doi: 10.1213/ANE.0000000000004517. PMID 31725024
- [Background] James PA, Oparil S, Carter BL, Cushman WC, Dennison-Himmelfarb C, Handler J, Lackland DT, LeFevre ML, MacKenzie TD, Ogedegbe O, Smith SC Jr, Svetkey LP, Taler SJ, Townsend RR, Wright JT Jr, Narva AS, Ortiz E. 2014 evidence-based guideline for the management of high blood pressure in adults: report from the panel members appointed to the Eighth Joint National Committee (JNC 8). JAMA. 2014 Feb 5;311(5):507-20. doi: 10.1001/jama.2013.284427. PMID 24352797
- [Background] Kim HY, Lee JE, Kim HY, Kim J. Volatile sedation in the intensive care unit: A systematic review and meta-analysis. Medicine (Baltimore). 2017 Dec;96(49):e8976. doi: 10.1097/MD.0000000000008976. PMID 29245269